CLINICAL TRIAL: NCT03462810
Title: GSK1265744 (Cabotegravir, CAB) for Named Patient/Compassionate Use in HIV
Status: Available | Type: Expanded Access
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 205741
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2020-10

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: cabotegravir, CAB; GSK1265744; Individual Patient Compassionate Use; HIV
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: cabotegravir, CAB — open label investigational product
  Other Names: cabotegravir; CAB

SUMMARY:
The goal of this compassionate use program is to provide a mechanism to supply Cabotegravir, CAB on an individual named patient basis for treatment of individuals who have no available treatment alternatives and/or limited treatment options (e.g., who are unable to participate in the Phase III clinical studies or do not qualify), and are in need of new drugs to construct an effective antiviral regimen and may require the use of parenterally administered drug given underlying medical conditions. You can access ViiV's Policy on Compassionate via https://us.viivhealthcare.com/media/124424/viivs-external-policy-on-cup_final-version_23feb2017.pdf.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients will be eligible for treatment if ALL the following apply:

  * Male or female patients aged ≥ 18 yrs

NOTE: all female patients of reproductive potential should use every precaution to prevent pregnancy including either complete abstinence from intercourse from 2 weeks prior to administration of CAB, throughout receipt of CAB and for at least 52 weeks after discontinuation of CAB LA; or use of one of the following methods of highly reliable contraception:

1. Contraceptive subdermal implant
2. Intrauterine device or intrauterine system
3. Combined estrogen and progestogen oral contraceptive
4. Injectable progestogen
5. Contraceptive vaginal ring
6. Percutaneous contraceptive patches
7. Male partner sterilisation with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. The documentation on male sterility can come from the site personnel's: review of subject's medical records, medical examination and/or semen analysis, or medical history interview provided by her or her partner.

These allowed methods of contraception are only effective when used consistently/correctly and in accordance with the product label. The investigator is responsible for ensuring that patients understand how to properly use these methods of contraception.

* Inability to construct a viable antiviral treatment regimen with commercially available medications;
* Demonstrated need for a long acting, injectable antiretroviral including, but not limited to malabsorption or inability to achieve adequate drug levels via oral route. NOTE: Poor/incomplete adherence to oral meds is not a sufficient rationale for inclusion.
* The patient/legal guardian or representative has given informed consent to treatment prior to administering CAB (in a manner consistent with all national requirements). The patient/legal guardian or representative has also given informed consent for the transmission of a copy of the anonymized adverse and serious adverse event (SAE) and pregnancy reports (in compliance with local regulatory authority requirements) to GSK and ViiV where allowable by local regulations, and to the country regulatory authority as required.

Exclusion Criteria:

* Patients will not be eligible for treatment if ANY of the following apply:

  * Patient has estimated creatinine clearance <50 mL/min via Cockcroft-Gault method;
  * Females who are pregnant or women who are breastfeeding, or plan to become pregnant or breastfeed during treatment.
  * Patients who have had known or suspected allergic reaction or hypersensitivity reactions to integrase inhibitors;
  * Alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN)
  * ALT ≥ 3 times ULN and bilirubin ≥ 1.5 times ULN (with > 35% direct bilirubin)
  * Evidence for moderate to severe hepatic impairment, grade 3-4 liver fibrosis, or cirrhosis
  * Patients who are eligible for actively enrolling clinical trials involving CAB.
  * Significant coagulopathy precluding chronic IM dosing

NOTE: Patients should not be treated via the named patient/compassionate use program if they are eligible and/or able to participate in any of the Phase III clinical trials of CAB and the patient is suitable for participation in such clinical trials. In that instance (assuming consent is obtained) the patient should preferentially be enrolled into the ongoing clinical trial to allow detailed data collection. In accordance with national requirements patients should not be treated in the named patient/compassionate use program if they have responded to previous treatment with CAB in another clinical trial without review and prior approval by the VSLC.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare